CLINICAL TRIAL: NCT02189135
Title: Making Ramadhan Fasting a Safer Experience With Technology Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Segi University (Other)
Responsible Party: Principal Investigator, Shaun Lee Wen Huey, Shaun Lee, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRFAST
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Usual care from physician/ doctor
- Telemedicine (Experimental): Mobile wireless glucometer with feedback from physicians
  Interventions: Device: Telemedicine

INTERVENTIONS:
Device: Telemedicine — The glucometer acts by automatically uploading any glucose readings to an online portal. A summary of the patient's glycaemic and metabolic control, self-management skills as well as compliance to other key measures such as eye examination, screening for microvascular complications would also be provided if available. All patients in this intervention arm would be given a system-driven guidance on when to test their blood glucose based on their disease status, medication regimen, and time of poorest control so that the most useful, patient specific blood profile can be created and used for future self-management coaching for patient
  Other Names: Myglucohealth wireless bluetooth glucometer
  Arms: Telemedicine

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a chronic condition that is one of the major causes of illness, disability, and death in Malaysia with an increasing prevalence. Despite the best effort, only 1 in 3 patients ever meet their HbA1c goal. In most patients with type 2 diabetes, the use of oral anti-diabetics is a mainstay in therapy. However, there is a risk of hypoglycaemia in most patients taking these drugs. This is especially important in T2DM Muslims wishing to fast during Ramadan as the dietary pattern changes to one large meal at sunset called 'Iftaar' and a light meal before dawn called 'Sahur'. Most Muslims will generally consume large quantities of fried and sugary foods when they break their fast or during the night. Given the importance and public health significance of poor diabetes management and its associated risk especially during Ramadan, the investigators aim to test the intervention of using remote monitoring within community provider practice for patients with T2DM. The investigators hypothesize that the combined use of a mobile enable glucometer which can directly feedback the patients glycaemic levels to the physicians will reduce and even eliminate the occurrence of hypoglycaemia whilst ensuring that patients remain euglycaemic throughout the whole Ramadan month.

DETAILED DESCRIPTION:
Eligible participants will be assigned based upon their participating site. Treatment assignments are unmasked. Intervention group will utilize a web enabled glucometer manufactured by Entra Health System (San Diego, California). The glucometer acts by automatically uploading any glucose readings to an online portal currently managed by Entra Health System. The web portal would host the patient's raw blood glucose in a logbook form and laboratory data. A summary of the patient's gylcaemic and metabolic control (lipid, blood pressure, weight) control, self-management skills as well as compliance to other key measures such as eye examination, screening for microvascular complications would also be provided if available. All patients in this intervention arm would be given a system-driven guidance on when to test their blood glucose based on their disease status, medication regimen, and time of poorest control so that the most useful, patient specific blood profile can be created and used for future self-management coaching for patient.

In the event that there is 3 continuous readings of hypoglycaemia (3.9mmol/L and below) or hyperglycaemia (11.1mmol/L and above), the system will automatically generate a message to inform the attending physician. The physician then has an option to use this information, but will remain responsible for all treatment decisions. For quality assurance, the physicians will be required to periodically review the participant's electronic logbook data and summary analysis reports, generated for patients and physicians. These feedbacks will be entered into an electronic logbook and captured real-time. A report will be generated summarizing the self-management actions for improving their diabetes control will be sent to the patients, physicians as well as family member every month. Each patient will also be informed that action plan serves as a pre-visit summary for the patient's next visit to their physician. In addition, the participant's family member(s) will also be invited to participate and if consented updated on the status of the participants blood glucose status periodically and be prompted whenever their glycaemic levels are beyond the target.

Participants assigned to the control group will continue to receive their usual medical care as they would from their physician or general practitioner including checking patient self-management blood glucose and log books. In addition, participants will receive standard lifestyle advice and will be given basic information on diabetes prevention, weight loss, diet, and exercise consistent with expert recommendation for a healthy lifestyle. Participants will also receive a glucose meter and supplies for 3 months. Participants will be told to use the glucose meter as recommended by their physicians. Control participants will also receive publically available literatures such as flyers and brochures.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed by a physician at least six months prior to study enrollment. This will be determined via self-report with verification (medical records, current treatment, or test results meeting the 2009 Malaysian Clinical Practice Guideline for Management of Type 2 Diabetes Mellitus (4th edition) criteria of fasting blood glucose > 7.0 mmol/L , symptoms of hyperglycaemia with casual plasma glucose >11.1mmol/L or two-hour plasma glucose >11.1mmol/L after a 75gram oral glucose load)
* HbA1c of > 7.5% but less than 11.0% within the most recent 3 months. Individuals with HbA1c exceeding this level may require more urgent care and as such will be asked to seek treatment
* Aged 18 - 75 years are eligible. Participants older than 75 years of age are excluded due to the increased risk of competing mortality and potential safety concerns related to hypoglycaemia
* Willing or has an intention to fast for at least 15 days during Ramadan
* Access to internet and an e-mail address , or access to a smartphone with 3G services in the intervention group
* Not pregnant or history of heart diseases, serious illness, cancer diagnosis or any other conditions that can impede participation

Exclusion Criteria:

* Unable or unwilling to give informed consent or communicate with local study staff
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* Hospitalization for depression in past six months
* Plans to relocate to an area or travel plans that do not permit full participation in the study
* Lack of support from primary health care provider or family members
* History of bariatric surgery, small bowel resection, or extensive bowel resection
* Currently pregnant or nursing
* Cancer: requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer)
* Cardiovascular disease (heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within last three months, stroke or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in past six months)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with hypoglycaemia in usual care versus telemedicine during Ramadan | Week 4

SECONDARY OUTCOMES:
Mean change in fructosamine from start of Ramadan (day -1) to end of Ramadan (day 29) in usual care versus telemedicine | Week 4
Total number of hypoglycaemic rates in usual care versus telemedicine during Ramadan | Week 4
Total number of hypoglycaemic rates in usual care versus telemedicine from baseline to end of treatment | Week 12
Glycaemic control of patients measured with HbA1c in patients under usual care versus telemedicine from baseline to end of treatment | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Lee, PhD, Principal Investigator — Monash University
Locations (1):
- Klinik Kesihatan Pandamaran, Klang, Selangor, Malaysia

REFERENCES:
- [Derived] Lee SWH, Chen WS, Sellappans R, Md Sharif SB, Metzendorf MI, Lai NM. Interventions for people with type 2 diabetes mellitus fasting during Ramadan. Cochrane Database Syst Rev. 2023 Jul 12;7(7):CD013178. doi: 10.1002/14651858.CD013178.pub2. PMID 37435938
- [Derived] Lee JY, Wong CP, Tan CSS, Nasir NH, Lee SWH. Type 2 diabetes patient's perspective on Ramadan fasting: a qualitative study. BMJ Open Diabetes Res Care. 2017 May 8;5(1):e000365. doi: 10.1136/bmjdrc-2016-000365. eCollection 2017. PMID 28761651
- [Derived] Lee JY, Lee SW, Nasir NH, How S, Tan CS, Wong CP. Diabetes telemonitoring reduces the risk of hypoglycaemia during Ramadan: a pilot randomized controlled study. Diabet Med. 2015 Dec;32(12):1658-61. doi: 10.1111/dme.12836. Epub 2015 Jul 15. PMID 26103794